CLINICAL TRIAL: NCT05157282
Title: Spinal Cord Stimulation for Functional Recovery in Humans With Tetraplegia
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: B3715-R
Record Dates: First submitted 2021-11-24; First posted 2021-12-14 (Actual); Last update posted 2026-01-16 (Actual); Status verified 2026-01

CONDITIONS: Spinal Cord Injury
Keywords: Spinal Cord Injury; Motor Function; Reaching; Grasping; Hand Movement
MeSH Terms: conditions — Spinal Cord Injuries

STUDY DESIGN:
Intervention Model Description: Transcutaneous electrical spinal stimulation (TESS)
Who Masked: Participant
Masking Description: Participants will not know if they receive real or sham stimulation
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (3):
- Active TESS Group 1 (Active Comparator): Subjects with SCI and without SCI (controls) will participate in two testing sessions, separated by 2-3 days, using a crossover design. In each session, active transcutaneous electrical spinal stimulation (TESS) will be applied over the cervical spinal cord. Functional and physiological measures will be acquired before and after each session.
  Interventions: Device: TESS; Other: Motor Task; Device: sham-TESS
- Sham TESS Group 1 (Sham Comparator): Subjects with SCI and without SCI (controls) will participate in two testing sessions, separated by 2-3 days, using a crossover design. In each session, sham transcutaneous electrical spinal stimulation (sham-TESS) will be applied over the cervical spinal cord. Functional and physiological measures will be acquired before and after each session.
  Interventions: Device: TESS; Other: Motor Task; Device: sham-TESS
- Active TESS + Training (Active Comparator): Develop methodologies to promote recovery of reaching and grasping movements. To accomplish this goal, the investigators will combine TESS applied in a closed-loop manner with massed practice upper-limb training. Participants will be assigned to one of three groups in a randomized order for a controlled design: [1) Closed-loop TESS applied during grasping + training, 2) Closed-loop TESS applied during reaching + training, and 3) Closed-loop TESS applied during grasping & reaching + training.] TESS for 20-min will be followed by 60 min of massed practice exercise training (total=20 sessions).
  Interventions: Device: TESS; Other: Training; Other: Motor Task

INTERVENTIONS:
Device: TESS — Small stimulation pulses will be given to the spine at C5-6 in a non invasive manner.
  Other Names: NeoStim-5
Other: Training — The participant will be instructed to do repetitive motor movements with their arm or hand.
  Other Names: Massed Practice Training
  Arms: Active TESS + Training
Other: Motor Task — Participants will be asked to perform specific motor tasks or movements with their fingers, hands, and arms.
Device: sham-TESS — Small sham stimulation pulses will be given to the spine at C5-6 in a non invasive manner.
  Other Names: NeoStim-5
  Arms: Active TESS Group 1; Sham TESS Group 1

SUMMARY:
In support of the long-term goal of developing new strategies to increase limb function after SCI, the objectives of this proposal are to: 1) Examine the behavioral and physiological effects of TESS on upper-limb muscles after cervical SCI; and 2) Maximize the recovery of reaching and grasping potential by using tailored TESS in a task-specific manner with motor training. Veterans with cervical spinal injuries and healthy volunteers will be recruited for this study.

DETAILED DESCRIPTION:
Current studies demonstrate that electrical spinal stimulation, either invasive or noninvasive, can play an important role in rehabilitation strategies aimed at improving limb function in humans with SCI (Taccola et al., 2018). Among current stimulation strategies, one of the most promising candidates to emerge in recent years is transcutaneous electrical spinal stimulation (TESS). TESS is a noninvasive technique that can be tailored to the needs of each individual, where several segments of the spinal cord can be stimulated at the same time, and delivery can be programed to interact with a rehabilitation strategy during functional movements, such as reaching or grasping. A key element to TESS is its ability to access spared spinal cord networks with minimal discomfort. Although promising, the knowledge of TESS remains limited in scope and more studies are needed to further identify its efficacy.

In Aim 1, subjects will participate in two randomized sessions: 1) TESS, and 2) sham-TESS.] In Aim 2, the investigators will examine the effect of stimulation and training for a total of 20 sessions (3 to 5 per week). Participants will be randomly assigned to: [1) Closed-loop TESS applied during grasping + training, or 2) Closed-loop TESS applied during reaching + training.]

AIM 1 Subjects with SCI and without SCI (controls) will participate in two testing sessions, separated by 2-3 days, using a crossover design. In each session, TESS or sham-TESS will be applied over the cervical spinal cord. Functional and physiological measures will be acquired before and after each session.

AIM 2 Develop methodologies to promote recovery of reaching and grasping movements. To accomplish this goal, the investigators will combine TESS applied in a closed-loop manner with massed practice upper-limb training. Participants will be assigned to one of three groups in a randomized order using a sham controlled design: [1) Closed-loop TESS applied during grasping + training, 2) Closed-loop TESS applied during reaching + training, and 3) Closed-loop TESS applied during grasping & reaching + training.] TESS for 20-min will be followed by 60 min of massed practice exercise training (total=20 sessions).

ELIGIBILITY:
Inclusion Criteria:

Inclusion criteria for SCI:

* Male and female Veterans between 18-70 years
* Chronic SCI (1 year of injury)
* Cervical injury at C8 or above - damage between cervical spinal segments will be confirmed using MRI [preliminary data (Benavides et al., 2020) and analysis of MRIs in ~100 participants with cervical SCI confirm that the investigators can meet our recruitment goals. Note that most SCI in humans damage several spinal cord segments

  * Verification of damage to cervical spinal segments will ensure that TESS electrodes will target the injured spinal cord (Benavides et al., 2020)
* Intact or impaired, but not absent, innervations in dermatomes C6, C7 and C8 during light touch and pin prick stimulus using the International Standards for Neurological Classification of Spinal Cord Injury (ISNCSCI) sensory scores as tested before in our studies (Bunday and Perez, 2012; Bunday et al., 2018; Benavides et al., 2020; Jo and Perez, 2020)
* Able to produce a visible power grip with one hand
* Can score a minimum of two (2) in the cylindrical grasp the "Prehension Ability" GRASSP

  * This criterion was selected to ensure that hand impairment will not interfere with the ability to perform training and the proposed tests

Inclusion criteria for controls:

* Males and females (18-70 years)
* Right-handed
* Able to complete grasping

Exclusion Criteria:

Exclusion criteria for SCI and control subjects:

* Uncontrolled medical problems including pulmonary, cardiovascular or orthopedic disease
* Any debilitating disease prior to the SCI that caused exercise intolerance
* Premorbid, ongoing major depression or psychosis, altered cognitive status
* History of head injury or concussion, skull fractures (or any skull deficit), unexplained headaches in the last 6 months, or stroke
* Pacemaker
* Metal plate in skull
* History of seizures
* Receiving drugs acting primarily on the central nervous system, which lower the seizure threshold, such as antipsychotic drugs (chlorpromazine, clozapine) or tricyclic antidepressants
* Pregnant females
* Ongoing cord compression, or a syrinx in the spinal cord, or one who suffers from a spinal cord disease such as spinal stenosis, spina bifida, or herniated cervical disk

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 86 (Estimated)
Dates: Start 2023-01-25 (Actual); Primary Completion 2027-01-29 (Estimated); Study Completion 2027-02-01 (Estimated)

PRIMARY OUTCOMES:
Changes in amplitude of Motor evoked potential size | Change from baseline at study completion, average of 5 weeks
  Ten stimuli (0.2 Hz) will be delivered at each intensity to plot the mean peak-to-peak amplitude of the MEP from the non-rectified response against the TMS intensity in each subject (MEP recruitment curve).
Change in GRASSP Test | Through study completion(average of 5 weeks) and during 6-month follow-up
  The GRASSP will be used to asses several domains of arm/hand function in humans with cervical SCI, specifically assessing three domains of hand function: 1) strength, 2) sensibility, and 3) prehension. The time to administer the test is ~45 min. The GRASSP has 5 subsets:
  * Dorsal sensation: (3 locations, each scored 0-4, sum=0-12)
  * Palmar sensation: (3 locations, each scored 0-4, sum=0-12)
  * Strength: (10 muscles of arm and hand, motor score 0-5, sum=0-50)
  * Prehension ability: (3 grasps (cylindrical, lateral key, tip to tip), each scored 0-4, sum=0-12)
  * Prehension performance: There are 6 prehension tasks. Pouring water from a bottle, opening jars, picking up and turning a key, transferring 9 pegs from board to board, picking up four coins and place in slots, screwing four nuts onto bolts. Each task is scored 0-5, sum=0-30.
Changes in amplitude of cervicomedullary motor evoked potential size | Change from baseline at study completion, average of 5 weeks
  Ten Transcranial magnetic stimuli (TMS) will be delivered to plot the mean peak-to-peak amplitude of the motor and cervicomedullary evoked potentials (MEPs and CMEPs, respectively) from the non-rectified response against the TMS intensity in each subject (MEP/CMEP recruitment curves).

CONTACTS AND LOCATIONS:
Overall Officials: Monica A Perez, PhD, Principal Investigator — Edward Hines Jr. VA Hospital, Hines, IL
Locations (2):
- United States (2):
  - Shirley Ryan AbilityLab, Chicago, Illinois
  - Edward Hines Jr. VA Hospital, Hines, IL, Hines, Illinois

IPD SHARING:
Plan to Share IPD: No